CLINICAL TRIAL: NCT04140149
Title: Living With Hope: A Preliminary Investigation of a Novel, CBT-Based Psychoeducational Skills Class for Individuals With a Recent Suicide Attempt
Brief Title: Living With Hope: A Preliminary Investigation of a Skills Class
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Christine Henriksen, Assistant Professor, University of Manitoba
Other Study IDs: H2019:292
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation
Keywords: Suicide; Suicide Attempt; Suicidal Ideation; Pilot; Intervention
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: Adults who have made a suicide attempt in the past 3 months who have been referred to, and enrolled in, the Living with Hope class.
  Interventions: Behavioral: Living with Hope

INTERVENTIONS:
Behavioral: Living with Hope — 12-week, CBT-based, psychoeducational skills class

SUMMARY:
This study will determine whether Living with Hope, a novel, 12-week coping skills class, reduces suicidal thoughts and behaviors among individuals who have made a recent suicide attempt. It is hypothesized that participants who complete the class will show significant improvements on measures of suicidal thoughts, hopelessness, and related mental health symptoms, and these improvements will be maintained over time.

DETAILED DESCRIPTION:
As the 9th leading cause of death worldwide, suicide is a major public health concern. One of the groups as highest risk of death are those that have previously made a suicide attempt. Effective treatment following a suicide attempt is imperative for reducing the risk of suicide, with increasing evidence showing treatments that target suicide behavior are more effective at reducing risk over treatments that target related mental health difficulties (e.g., depression). However, these treatments are resource intensive and are difficult to access in Manitoba, and many individuals who have made a suicide attempt do not receive any mental health treatment. In order to ensure timely access to treatment following a suicide attempt, we have created a non-resource intensive psychoeducational skills class grounded in evidence-based suicide-specific treatment. The primary aim of this study is to examine the safety and effectiveness of a novel, 12-week cognitive behavior therapy-based, virtual psychoeducational skills class (Living with Hope) in reducing suicidal thoughts and behaviors among adults who have made a recent suicide attempt, and determine whether changes post-treatment are maintained at over time. The secondary aim is to determine whether this intervention also results in improvements on related mental health outcomes, and whether changes on these constructs mediate improvements on suicidal thoughts and behaviors.

Adults ages 18 years and older who have been referred to the Living with Hope class over the 2 year study period will be invited to participate in the proposed study (anticipated n=60). Individuals are eligible for referral if they have made a suicide attempt in the past 3 months and are either seeking mental health crisis services. Participants will complete standardized measures of primary (suicidal thoughts and behaviors) and secondary outcomes (hopelessness, depressive symptoms, emotion regulation difficulties, and quality of life) at pre-treatment, mid-way through the 12-week class, post-treatment, 1-month follow-up, and 3-months follow-up. Mixed-effects linear regression will determine whether there are significant differences on outcome measures at any of these five time-points, as well as whether secondary outcomes mediate improvements on primary outcomes. All research participation will be conducted through virtual means.

The proposed study would be the first in Canada to examine the effectiveness of a low-cost, targeted psychoeducational skills class in reducing suicidal thoughts and behaviors among individuals who have made a recent suicide attempt. This will set the stage for future linkage with administrative data and randomized controlled trials aimed at determining whether the Living with Hope class results in reduced suicide attempts and deaths compared to treatment as usual. If proven safe and effective through these rigorous evaluations, the Living with Hope class could be widely disseminated in the public health system to provide care to a large number of Manitobans, with the long-term goal of increasing access to timely, targeted treatment, and in turn, reducing suicides in Manitoba.

ELIGIBILITY:
Inclusion Criteria:

1. Made a suicide attempt in the past 3 months
2. Sought mental health crisis services, and referred to the Living with Hope program

   -

Exclusion Criteria:

1. Not proficient in English
2. Exhibiting active psychotic symptoms
3. Significant cognitive impairment, are
4. Currently expressing anger or disappointment about the outcome of their attempt,
5. Recent history of violence or verbal aggression towards others, or are exhibiting other signs of behavior that would pose a threat to the safety or wellbeing of class participants 6. Primary substance use disorder -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 years and older who have made a suicide attempt in the past 3 months and have sought mental health help through a local crisis response centre or emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Beck Scale for Suicide Ideation | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  21 item self-report measure of the severity of past-week suicidal ideation
Change in scores on the Columbia-Suicide Severity Rating Scale | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  Clinician-administered interview schedule designed to measure the timing and frequency of suicidal thoughts and behaviors
Suicide attempts | Through the duration of treatment and over follow-up period (approximately 6 months)
  Presence of a suicide attempt during the study or over the follow-up period, as assessed by the Columbia-Suicide Severity Rating Scale

SECONDARY OUTCOMES:
Change in scores on The Beck Hopelessness Scale | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  20-item self-report measure of past-week hopelessness and negative beliefs about the future
Change in scores on the Patient Health Questionnaire-9 | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  9-item self-report measure of depressive symptom severity over the past two-weeks
Change in scores on the Difficulties in Emotion Regulation Scale | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  36-item measure of current emotional dysregulation difficulties
Change in scores on the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Change from baseline to mid-treatment (approximately 7 weeks), to post-treatment (approximately 14 weeks), to 1-month follow-up, and to 3-month follow-up
  16-item self-report measure of current quality of life
Safety Item | Week 1 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 2 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 3 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 4 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 5 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 6 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 7 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 8 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 9 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 10 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 11 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings
Safety Item | Week 12 of Living with Hope class session
  One item assessing the degree that the Living with Hope class session increased a participant's suicidal feelings

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Henriksen, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Crisis Response Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The research team has not determined whether de-identified individual participant data will be made available to other researchers after the completion of this study, as it is unclear whether our institution has a separate ethical approval process for this and what the requirements for this would be, if so. Additionally, it is unclear whether there is established infrastructure to ensure data are securely transferred to any potentially interested researcher to protect participants.